CLINICAL TRIAL: NCT04383899
Title: Role of Ibuprofen and Other Medicines on Severity of Coronavirus Disease 2019 (COVID-19) Infections: a Case-control Study
Brief Title: Role of Ibuprofen and Other Medicines on Severity of Coronavirus Disease 2019
Acronym: RISC
Status: Withdrawn | Type: Observational
Why Stopped: Ibuprofen is not prescribed during coronavirus pandemic, so the study is stopped
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux PharmacoEpi (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/13
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection
Keywords: NSAID; Ibuprofen; chronic pathology
MeSH Terms: conditions — Coronavirus Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patient: Patients from the cohort with severe coronavirus infection necessitating intensive care (artificial ventilation) with ulterior recovery or fatal outcome.
  Interventions: Other: Questionnaire
- Control patient: All patients from the cohort with non-severe coronavirus infection, who were not admitted to hospital or who were admitted to hospital but without the need for intensive care, and who recovered.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — All patients testing positively for COVID-19, with completed questionnaires. As appropriate, the duration of the study will be at least the time to complete the questionnaire for non-hospitalized patients, and for those who are hospitalized, they will be followed until hospital discharge or death to ascertain outcome.

SUMMARY:
It has been suggested that ibuprofen might be associated with more severe cases of coronavirus infections, based on the observation that severe COVID cases had been exposed to ibuprofen, resulting in a warning by the French authorities.

This was attributed to:

1. a suggestion that ibuprofen might upregulate ACE-2 thereby increasing the entrance of COVID-19 into the cells,
2. an analogy with bacterial soft-tissue infections where more severe infections on NSAIDs are attributed to an immune-depressive action of NSAIDs, or to belated treatment because of initial symptom suppression,
3. fever is a natural response to viral infection, and reduces virus activity: antipyretic activity might reduce natural defenses against viruses. However fever reduction in critically ill patients had no effect on survival.

However, these assertions are unclear: upregulation of ACEII would increase the risk of infection, not necessarily its severity, and would only apply to the use of NSAIDs before the infection, i.e. chronic exposure. It would be irrelevant to the infection once the patients are infected, i.e., to symptomatic treatment of COVID-19 infection.

Anti-inflammatory effect masking the early symptoms of bacterial infections resulting in later antibiotic or other treatment is not applicable: there is no treatment of the virus that might be affected by masking symptoms.

Antipyretic effect increasing the risk or the severity of infection would apply equally to all antipyretic agents including paracetamol, which share the same mechanism of action for fever reduction.

EMA remains prudent about this assertion

In addition, excess reliance on paracetamol while discouraging the use of ibuprofen might increase the risk of hepatic injury from paracetamol overdose. Paracetamol is the prime drug associated with liver injury and transplantation, in voluntary and inadvertent overdose or even at normal doses. This might be increased by COVID-related liver function alterations.

It is therefore proposed to conduct a case-control study in a cohort of patients admitted to hospital in France with COVID-19 infection.

DETAILED DESCRIPTION:
It has been suggested that ibuprofen might be associated with more severe cases of coronavirus infections, based on the observation that severe COVID cases had been exposed to ibuprofen, resulting in a warning by the French authorities (published in a french journal called "Le Monde" = The world).

This was attributed to:

1. a suggestion that ibuprofen might upregulate ACE-2 thereby increasing the entrance of COVID-19 into the cells.This is based on a single study in streptozotocin-induced diabetic rats where ibuprofen decreases cardiac fibrosis. There seems to be no study in man. (https://www.dw.com/en/coronavirus-confusion-about-safety-of-ibuprofen/a-52824043) These authors noted an increased risk of severe COVID-19 in patients with hypertension or diabetes, and a possible role of Angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) which also upregulate ACE-2, as do also thiazolidinedione antidiabetic drugs. The relevance of this up-regulation seems disputed.
2. an analogy with bacterial soft-tissue infections where more severe infections on NSAIDs are attributed to an immune-depressive action of NSAIDs, or to belated treatment because of initial symptom suppression.
3. fever is a natural response to viral infection, and reduces virus activity: antipyretic activity might reduce natural defenses against viruses. However fever reduction in critically ill patients had no effect on survival. A meta-analysis of fever reduction in children found no difference on outcomes between paracetamol and ibuprofen.

However, these assertions are unclear: upregulation of ACEII would increase the risk of infection, not necessarily its severity, and would only apply to the use of NSAIDs before the infection, i.e. chronic exposure. It would be irrelevant to the infection once the patients are infected, i.e., to symptomatic treatment of COVID-19 infection.

Anti-inflammatory effect masking the early symptoms of bacterial infections resulting in later antibiotic or other treatment is not applicable: there is no treatment of the virus that might be affected by masking symptoms.

Antipyretic effect increasing the risk or the severity of infection would apply equally to all antipyretic agents including paracetamol, which share the same mechanism of action for fever reduction.

EMA remains prudent about this assertion (EMA gives advice on the use of non-steroidal anti-inflammatory drugs for COVID-19, 18 March 2020 EMA/136850/2020).

These findings raise the question of

1. an indication bias, where more severe cases with more symptoms and higher fever might not respond well to the first line antipyretic paracetamol, so that ibuprofen was then used. (reverse causality) The same has been described with soft-tissue infection
2. the reality of an increased risk in patients chronically on drugs that upregulate ACEII, such as NSAIDs, antihypertensive drugs and especially ACEI or ARB, or antidiabetic drugs and especially thiazolidinediones.
3. the impact of concomitant or pre-existing diseases such as diabetes, hypertension or heart failure.

In addition, excess reliance on paracetamol while discouraging the use of ibuprofen might increase the risk of hepatic injury from paracetamol overdose. Paracetamol is the prime drug associated with liver injury and transplantation, in voluntary and inadvertent overdose or even at normal doses. This might be increased by COVID-related liver function alterations.

It is therefore proposed to conduct a case-control study in a cohort of patients admitted to hospital in France with COVID-19 infection, to explore these different questions.

ELIGIBILITY:
Inclusion Criteria:

- All patients tested for COVID-19 in hospital centers participating to the study.

No exclusion Criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be screened at the time of their visit to the participating hospital center; i.e. at the ambulatory screening center adjacent to the hospital not necessarily resulting in patient hospitalization, or directly on admission at the appropriate hospital department (emergencies, intensive care or others).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Describe medications used prior to admission associated with worse infection in COVID-19 patients in France. | At inclusion day
  Describe medications including ibuprofen used prior to admission associated with worse infection in COVID-19 patients in France. Thanks to a questionnaire created for the study, with 5 questions on existing pathology, drugs administrated symptom onset and when, hospitalisation. Each questions have a multiple choice.
Quantify medications used prior to admission associated with worse infection in COVID-19 patients in France. | At inclusion day
  Quantify medications including ibuprofen used prior to admission associated with worse infection in COVID-19 patients in France. Thanks to a questionnaire created for the study, with 5 questions: existing pathology, drugs administrated symptoms onset and when, hospitalisation. Each questions have a multiple choice.

SECONDARY OUTCOMES:
Describe other patient characteristics with worse infection in COVID-19 patients in France. | At inclusion day
  Describe patient characteristics thanks to the same questionnaire.
Quantify other patient characteristics with worse infection in COVID-19 patients in France. | At inclusion day
  Quantify patient characteristics thanks to the same questionnaire.

IPD SHARING:
Plan to Share IPD: No